CLINICAL TRIAL: NCT04436250
Title: Intravenous Infusions of S-KETAMINE in Fibromyalgia Syndromes: an Exploratory Study.
Brief Title: ESKETamine for FIBromyalgia Treatment
Acronym: ESKEFIB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ESKEFIB
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 2:1 ratio (S-ketamine : placebo) per block of 15 patients sequentially into the first 2 groups, one with placebo and one with first dose of S-Ketamine Low Dose (0.2mg/kg).
  A second group will receive S-Ketamine High Dose (0.4 mg/kg) with the same randomized ratio (2:1).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research pharmacist prepares the syringe with a placebo or active drug (group 1 with 0.2mg/kg or group 2 with 0.4 mg/kg of S-Ketamine) and anonymizes it before giving it to care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Active Comparator): Clonidine at a dose of 1 microg/kg Magnesium sulfate at a dose of 40 mg/kg
  Interventions: Drug: Active comparator
- S-Ketamine Low dose (Experimental): S-Ketamine at a dose of 0.2 mg/kg
  Interventions: Drug: Active comparator; Drug: S-Ketamine Low dose
- S-ketamine High dose (Experimental): S-ketamine at a dose of 0.4 mg/kg
  Interventions: Drug: Active comparator; Drug: S-Ketamine High dose

INTERVENTIONS:
Drug: Active comparator — The active comparator is composed of clonidine 1 microg/kg combined with magnesium sulfate 40 mg/kg diluted in 45 ml of sodium chloride
Drug: S-Ketamine Low dose — The arm 1 is composed of esketamine 0.2 mg/kg and clonidine 1 microg/kg combined with magnesium sulfate 40 mg/kg diluted in 45 ml of sodium chloride.
  Arms: S-Ketamine Low dose
Drug: S-Ketamine High dose — The arm 2 is composed of esketamine 0.4 mg/kg and clonidine 1 microg/kg combined with magnesium sulfate 40 mg/kg diluted in 45 ml of sodium chloride.
  Arms: S-ketamine High dose

SUMMARY:
Fibromyalgia is a cause of chronic pain, classified by the Internal Classification of Diseases (ICD) as a primary chronic pain with specific diagnostic criteria established by the American College of Rheumatology (ACR). No treatment to its complete cure is available at this time, all treatments having as purpose pain relief and an improvement of quality of life by combining pharmacologic and nonpharmacologic treatments. One of the mechanisms proposed in fibromyalgia is the central sensitisation phenomenon, by which the central nervous system becomes "hypersensitive" to nociceptive or non-nociceptive stimuli. The receptor involved in this phenomenon is the N-methyl-D-aspartate receptor to which ketamine binds. Ketamine has therefore been proposed as a co-treatment in chronic pain with central sensitization phenomena, such as fibromyalgia.

DETAILED DESCRIPTION:
Ketamine is a drug used for anesthesia since the 1970s, acting as an antagonist to the N-methyl-D-aspartate receptor located in the central nervous system. It has two stereoisomers : R +ketamine and S - ketamine, the latter being about two to four times more potent. S-ketamine also has the advantages of producing less psychotropic effects, less tiredness and a lower temporary cognitive impairment than the racemic mixture at equianalgesic doses. Being first used as an anesthetic, in the last twenty years, ketamine's indications expanded to other domains, such as treatment of depression or off label use for chronic pain relief. Chronic pain is a multidimensional syndrome that touches 17-44% of the population of western countries. Fibromyalgia is a cause of chronic pain, classified by the Internal Classification of Diseases (ICD) as a primary chronic pain with specific diagnostic criteria established by the American College of Rheumatology (ACR). No treatment to its complete cure is available at this time, all treatments having as purpose pain relief and an improvement of quality of life by combining pharmacologic and nonpharmacologic treatments (as given by the European League Against Rheumatism (EULAR) guidelines). One of the mechanisms proposed in fibromyalgia is the central sensitisation phenomenon, by which the central nervous system becomes "hypersensitive" to nociceptive or non-nociceptive stimuli. The receptor involved in this phenomenon is the N-methyl-D-aspartate receptor to which ketamine binds. Ketamine has therefore been proposed as a co-treatment in chronic pain with central sensitization phenomena, such as fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from chronic pain (as defined by International Association for the Study of Pain) being diagnosed as fibromyalgia according to the American College of Rheumatology 2016 criteria
* patients qualified for the treatment by S-ketamine as established by our latest clinical practice
* patients aged 18-65 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is twofold, aiming on one side pain relief and on the other the improvement of the patient's functional status | 12 weeks
  Pain relief will be considered as a two point decrease on the Brief Pain Inventory (BPI) pain severity index at twelve weeks follow-up. (Two points being established as the Minimal Clinically Important Difference (MCID) for fibromyalgic patients).
  The functional status will be evaluated by the BPI Interference scale. An improvement will be considered as a one point reduction on this index (as established by the MCID).
  The primary outcome is to determine whether the association of S-ketamine to the analgesic treatment will increase the number of patients showing a clinically significant improvement of pain and/or functional status.

SECONDARY OUTCOMES:
Number of patients showing 50 % reduction in the BPI (Brief Pain Inventory) pain index | 12 weeks
  Measures will be done with different questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Lechat, MD, Principal Investigator — Grand Hôpital de Charleroi
Locations (1):
- Grand Hôpital de Charleroi, Gilly, Hainaut, Belgium

REFERENCES:
- [Derived] Javorcikova Z, Dangoisse M, Nikis S, Lechat JP, Gillain A, Fils JF, Van der Linden P. The place of S-ketamine in fibromyalgia treatment (ESKEFIB): study protocol for a prospective, single-center, double-blind, randomized, parallel-group, dose-escalation controlled trial. Trials. 2021 Nov 27;22(1):853. doi: 10.1186/s13063-021-05814-4. PMID 34838114